CLINICAL TRIAL: NCT05269030
Title: The Potential Therapeutic Effect of Ivermectin Nasal Drops in the Treatment of Post COVID-19 Parosmia
Brief Title: Ivermectin Nasal Drops in Post COVID-19 Parosmia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmad Mahmoud Hamdan, Principal Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2022 PHAR
Record Dates: First submitted 2022-03-04; First posted 2022-03-07 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Parosmia
Keywords: Ivermectin; Olfactory dysfunction; Parosmia; Post COVID-19 Parosmia
MeSH Terms: conditions — Olfaction Disorders | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to the patient's group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): The patients will receive ivermectin nasal drops
  Interventions: Drug: Ivermectin Topical
- Control group (Active Comparator): The patients will receive local steroid spray
  Interventions: Drug: Budesonide Nasal

INTERVENTIONS:
Drug: Ivermectin Topical — Ivermectin 1% in a dose of two drops per nostril twice daily.
  Arms: Case group
Drug: Budesonide Nasal — 64 µg per puff in a dose of 1 puff for each nostril twice daily.
  Arms: Control group

SUMMARY:
The current study will be a pilot study for a randomized controlled trial conducted on patients recruited from the outpatient clinic of the Otorhinolaryngology Department, Menoufia Faculty of Medicine To evaluate the effect of ivermectin nasal drops in the treatment of post COVID 19 parosmia

DETAILED DESCRIPTION:
The current study will be a pilot study for a randomized controlled trial conducted on 60 patients recruited from the outpatient clinic of the Otorhinolaryngology Department, Menoufia Faculty of Medicine after approval of the institutional review board and taking informed written consent from every patient before participation in the study.

To be included in the study, patients should be more than 18 years old, have a history of COVID 19 infection more than three months ago as confirmed by PCR test, have a post COpost-COVIDVID parosmia, and have no history of systemic steroid administration over the last one month. History of previous nasal surgery, underlying systemic diseases (like diabetes mellitus, hypertension, or autoimmune diseases), and hypersensitivity to Ivermectin were the exclusion criteria for this study.

Patients of the study will be randomly and equally distributed between case and control groups using block randomization methods using 4 blocks each comprising 4 patients with 6 patterns for every block one of which was selected randomly using random numbers generated by Excel program. Case group will receive a 4 weeks course of Ivermectin 1% in a dose of two drops per each nostril twice daily. Control group will receive a 4 weeks course of local steroids in the form of budesonide (64 µg per puff in a dose of 1 puff for each nostril twice daily.

Assessment protocol:

Patients of the study will be assessed before and at the end of the treatment protocol with history taking to define the inclusion and exclusion criteria. Endoscopic examination of the nasal cavity will be performed to exclude any other intranasal pathology. The degree of parosmia will be assessed using a visual analog scale before and four weeks after treatment.

Outcome measures:

Primary outcome measures will include a comparison between the pre and post treatment values of visual analog scales of parosmia, and a comparison between case and control groups regarding the post treatment results whether no improvement, partial improvement, or complete improvement. Secondary outcome measures will include assessment of the side effects of Ivermectin nasal drops among the case group.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be more than 18 years old,
* Patients having a history of COVID 19 infection more than three months ago as confirmed by PCR test,
* Patients having a post COVID parosmia,
* Patients having no history of systemic steroid administration over the last one month.

Exclusion Criteria:

* History of previous nasal surgery,
* Underlying systemic diseases (like diabetes mellitus, hypertension, or autoimmune diseases),
* Hypersensitivity to Ivermectin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between the pre and post treatment values | After one month of treatment
  Comparison between the pre and post-treatment values of visual analog scale values for post-COVD-19 parosmia. The values range from 0 to 10 with 10 indicating severe parosmia
Comparison between case and control groups regarding the post treatment results | After one month of treatment
  Comparison between case and control groups regarding the post treatment results whether no improvement, partial improvement, or complete improvement

SECONDARY OUTCOMES:
Assessment of the side effects of Ivermectin nasal drops | After one month of treatment
  Assessment of the side effects of Ivermectin nasal drops among the case group

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request from the authors
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of the study
Access Criteria: On approval of the authors

REFERENCES:
- [Background] Stenner M, Vent J, Huttenbrink KB, Hummel T, Damm M. Topical therapy in anosmia: relevance of steroid-responsiveness. Laryngoscope. 2008 Sep;118(9):1681-6. doi: 10.1097/MLG.0b013e31817c1368. PMID 18677278
- [Background] Butowt R, von Bartheld CS. Anosmia in COVID-19: Underlying Mechanisms and Assessment of an Olfactory Route to Brain Infection. Neuroscientist. 2021 Dec;27(6):582-603. doi: 10.1177/1073858420956905. Epub 2020 Sep 11. PMID 32914699
- [Background] Gane SB, Kelly C, Hopkins C. Isolated sudden onset anosmia in COVID-19 infection. A novel syndrome? Rhinology. 2020 Jun 1;58(3):299-301. doi: 10.4193/Rhin20.114. PMID 32240279
- [Background] Graziadei PP, Levine RR, Monti Graziadei GA. Plasticity of connections of the olfactory sensory neuron: regeneration into the forebrain following bulbectomy in the neonatal mouse. Neuroscience. 1979;4(6):713-27. doi: 10.1016/0306-4522(79)90002-2. No abstract available. PMID 481748
- [Background] Hornung DE, Mozell MM. Factors influencing the differential sorption of odorant molecules across the olfactory mucosa. J Gen Physiol. 1977 Mar;69(3):343 -61. doi: 10.1085/jgp.69.3.343. PMID 300427
- [Background] Conterno LO, Turchi MD, Correa I, Monteiro de Barros Almeida RA. Anthelmintic drugs for treating ascariasis. Cochrane Database Syst Rev. 2020 Apr 14;4(4):CD010599. doi: 10.1002/14651858.CD010599.pub2. PMID 32289194
- [Background] Kahlenberg JM, Kaplan MJ. Little peptide, big effects: the role of LL-37 in inflammation and autoimmune disease. J Immunol. 2013 Nov 15;191(10):4895-901. doi: 10.4049/jimmunol.1302005. PMID 24185823
- [Background] Heidary F, Gharebaghi R. Ivermectin: a systematic review from antiviral effects to COVID-19 complementary regimen. J Antibiot (Tokyo). 2020 Sep;73(9):593-602. doi: 10.1038/s41429-020-0336-z. Epub 2020 Jun 12. PMID 32533071
- [Background] Errecalde J, Lifschitz A, Vecchioli G, Ceballos L, Errecalde F, Ballent M, Marin G, Daniele M, Turic E, Spitzer E, Toneguzzo F, Gold S, Krolewiecki A, Alvarez L, Lanusse C. Safety and Pharmacokinetic Assessments of a Novel Ivermectin Nasal Spray Formulation in a Pig Model. J Pharm Sci. 2021 Jun;110(6):2501-2507. doi: 10.1016/j.xphs.2021.01.017. Epub 2021 Jan 23. PMID 33493479
- [Background] Aref ZF, Bazeed SEES, Hassan MH, Hassan AS, Rashad A, Hassan RG, Abdelmaksoud AA. Clinical, Biochemical and Molecular Evaluations of Ivermectin Mucoadhesive Nanosuspension Nasal Spray in Reducing Upper Respiratory Symptoms of Mild COVID-19. Int J Nanomedicine. 2021 Jun 15;16:4063-4072. doi: 10.2147/IJN.S313093. eCollection 2021. PMID 34163159